CLINICAL TRIAL: NCT01048489
Title: Effectiveness of a Community Integrated Program to Reduce Smoking Incidence in High School Students
Brief Title: Evaluation of a Program to Reduce Smoking in High School Students
Acronym: TAB_es
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Institut Catala de Salut (Other Government)
Responsible Party: Empar Valdivieso López, Institut Catala de Salut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI070937
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-12

CONDITIONS: Smoking in Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Other)
  Interventions: Behavioral: Health education in the high school
- No counseling (No Intervention)

INTERVENTIONS:
Behavioral: Health education in the high school — (12- 13 years old): 1.Questionnaire and measuring of carbon monoxide in air. 2.Role Games.3.Build a machine that simulates a cigarette.
  (13-14 years old):1.Questionnaire and measuring of carbon monoxide in air.2. Workshop dealing with current television series broadcast in Spain in which tobacco is constantly present.3.Workshop dedicated to make young people and their families stop smoking.A competition is performed between all the schools in order to reward the bookmark with the best motto asking any close person to stop smoking or thanking them for having quit.
  (14-15 years old):1.Questionnaire and measuring of carbon monoxide in air. 2. Workshop to go into depth about tobacco effects,by searching in the internet, aiming for the creation of an anti-tobacco pressure group in social networks such like Facebook.3.Workshop to create an advertising campaign to encourage non-consumption by mobile messages,use of internet..coinciding with the international day without tobacco.
  Arms: Lifestyle counseling

SUMMARY:
Effectiveness of health education regarding the smoking habit is under discussion . Nevertheless, according to the literature, some personal, familiar, cultural, and social factors are considered risk factors for students to become smokers. Probably, a health education intervention integrated in the school program will show a higher rate of effectiveness regarding incidence and prevalence of smoking habit in this age-group .

OBJECTIVE: To evaluate the effectiveness of a health education program to reduce the smoking habit in students.

METHODOLOGY: Quasi-experimental design including all the junior high school students in an educational district in Tarragona (Spain). The sampled schools will be randomised into two groups (experimental and control). All the included students will be monitored for three years.

The health education program will be divided in three interventions: role games and debates (1st year), workshops regarding the family and the social role of smoking (2nd year) , and the analysis of smoking advertising (3rd year). The incidence and prevalence rates will be compared on the experimental and control group, before de beginning of the intervention and at the beginning of each year.

ELIGIBILITY:
Inclusion Criteria:

* Students in high school
* Male and female
* Ages 12 to 16 years old

Exclusion Criteria:

* No Spanish speakers

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2256 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence of smoking is measured annually at the beginning and end of each school year by the use of a validated questionnaire and by the monitoring of carbon monoxide in expired air | January 2007 at June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Empar Valdivieso, RN, MSN, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Institut Català de la Salut, Tarragona, Tarragona, Spain

REFERENCES:
- [Background] Valdivieso López A, Ledo Garcia J, Barrera Uriarte M, Rivera Bosch G, Fuentes Bellido CM. Muniain Diaz de Cerio MP. Efectividad de un programa comunitario integrado en la escuela para reducir la incidencia de tabaquismo entre los escolares de ESO. Nure Investigación 2005;14. available at: http://www.fuden.es/proyectos_detalle.cfm?ID_INV_NURE=37&FilaInicio=21